CLINICAL TRIAL: NCT04050995
Title: Evaluating the Validity, Reliability, and Clinical Utility of the Music Therapy Sensory Instrument for Cognition, Consciousness and Awareness (MuSICCA) in Children and Youth With Prolonged Disorders of Consciousness
Brief Title: Evaluation of the MuSICCA for Measuring Awareness
Status: Recruiting | Type: Observational
Sponsor: The Children's Trust, United Kingdom (Other)
Collaborators: Temple University (Other)
Responsible Party: Sponsor
Other Study IDs: TCT 021; 167534 (Other: National Health Service Health Research Authority)
Record Dates: First submitted 2019-08-07; First posted 2019-08-09 (Actual); Last update posted 2025-04-30 (Actual); Status verified 2025-04

CONDITIONS: Disorder of Consciousness
MeSH Terms: conditions — Consciousness Disorders

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Weeks
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Prolonged Disorders Of Consciousness (PDOC) include the Vegetative State (VS) and the Minimally Conscious State (MCS) that persist for longer than four weeks. This research seeks to evaluate the validity (accuracy), reliability, and clinical utility (usefulness to clinicians) of the children's version of the Music Therapy Assessment Tool for Awareness in Disorders of Consciousness (MATADOC). The paediatric version is called the Music therapy Sensory Instrument for Cognition, Consciousness and Awareness (MuSICCA). The MATADOC is known to be accurate in diagnosis and has been shown to be clinically useful when working with adults. However, currently, there are no equivalent measures that have been rigorously tested for working with children. Therefore, there is a significant need for a valid and reliable measure, especially when the consequences of misdiagnosis include insufficient care provision, unsuitable treatment programmes, poor identification of intentions to communicate, and insufficient evidence for making difficult decisions around withdrawal of hydration and nutrition.

The study will invite participants aged 2-18 years, who the medical team suspect of having a PDOC, from various medical facilities in the UK, Ireland and other English-speaking countries. Parental/carer consent will be required for inclusion in the study.

Data collection will occur over 3 years. Each participant will be involved once for a maximum of 7 assessment sessions (4 for the MuSICCA, 1 for the Coma Recovery Scale - Revised (CRS-R), 1 for the Coma/Near Coma Scale (CNC), and 1 for the Nociception Coma Scale Revised (NCS-R)). The MuSICCA assessment protocol involves presenting musical stimuli in three modalities (visual, auditory, and tactile). The participants will be instructed to respond to stimuli and commands. Sessions will be recorded using audio-visual equipment and physical responses will be noted on documentation. The information gained will inform diagnosis and treatment. The participants' behaviours will also be scored on the CRS-R (the gold standard for diagnosis of DOC in adults), the CNC and the NCS-R.

DETAILED DESCRIPTION:
The null hypotheses are as follows:

The MuSICCA is not a valid tool for use with children and young people with Disorders Of Consciousness (DOC).

The MuSICCA is not a reliable tool for use with children and young people with DOC.

The MuSICCA is not a clinical useful tool for use with children and young people with DOC.

The design has been chosen to test the validity and reliability of the MuSICCA. It will involve carrying out the two measures and comparing their results against the current gold standard (the Coma Recovery Scale-Revised) and the Coma-Near Coma Scale. The design is influenced by previous validation studies of these measures conducted with adults.

There will be no control group because this is not a Randomised Controlled Trial (RCT) and, therefore, no recruited participant will be deprived of the potential benefits of the measures. All participants will receive intervention through the administration of the protocols of the assessment measures.

The study intends to recruit 80 participants. Recruitment will involve the following procedure. Medical/clinical teams at each site will identify potential participants according to the inclusion and exclusion criteria. The participants' families will be contacted to invite them to a meeting to discuss the research. It will be made clear that there will be no obligation to attend the meeting and their care or treatment will not be reduced or withdrawn if they decide not to be involved in the study. Interested families will be informed about the research project at this initial meeting. This information will be delivered verbally in person by the assessing clinicians and the families will be given a participant information sheet, which will contain all the information about the research so that the family can think in their own time about the decision to involve their child. The information given will include: 1)what will be carried out during the assessments, 2)how data will be recorded (observation recording sheets, video recording), 3)how the data will be stored, 4)what the data will be used for, and 5)what will be done with the data when the study has finished. The information sheet will also contain information about the families' right to withdraw their child from the study at any time without consequence.

The families will also be given the opportunity to ask questions so that they are satisfied that they understand why the research is being conducted, what the research will involve, and the extent of their child's involvement in the study if recruited.

Data collection will take place over a 3-year period at sites in the United Kingdom (UK), United States, and other English-speaking countries, e.g. Australia, Canada and New Zealand.

The data will consist of hand scored forms of the assessment tools and audio-visual recordings of the MuSICCA sessions. These recordings will be used to test the reliability of the MuSICCA between assessors and between assessment sessions.The selection and allocation of video recordings of sessions for inter-rater reliability will be carried out to control for differences of experience between assessing clinicians.

In order to eliminate researcher bias, data will be collated by the trained assessors from the treating clinical team, and statistical analysis will be undertaken by an independent statistician. In order to eliminate bias during data collection, there will be no interim data analysis and data collectors (clinicians) will not be able to discuss with each other the findings of their assessments until after the assessments have been completed and the results submitted to the research assistant.

Clinical utility of the MuSICCA will be evaluated using a questionnaire for each family and each assessing clinician using the tool. After each MuSICCA report is submitted and feedback given to the families, assessing clinicians and families will be asked to complete a short questionnaire to assess the clinical utility of the MuSICCA.

Data storage Raw data (score forms and video recordings) will be stored on a secure cloud-based system. Access to the data will be managed and authorised by the Chief Investigator.

Data analysis will be carried out by an independent statistician.

ELIGIBILITY:
Inclusion Criteria:

* Between 2-18 years of age
* Assessed by the interdisciplinary team as having a disorder of consciousness
* Be under active investigation for diagnosis of DOC

Exclusion Criteria:

* Known hearing impairments
* Known profound visual impairments
* Known musicogenic epilepsy
* Seizure disorders that cause frequent and/or prolonged seizures
* English not first language

Ages: 2 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Children and young people aged 2-18 years with a suspected disorder of consciousness. They will be identified by the treating clinical team initially.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2022-04-01 (Actual); Primary Completion 2026-12-01 (Estimated); Study Completion 2027-12-01 (Estimated)

PRIMARY OUTCOMES:
Music therapy Sensory Instrument for Cognition, Consciousness and Awareness | 2 weeks
  Measure of awareness
Coma Recovery Scale - Revised | 1 day
  Diagnostic tool for disorders of consciousness

SECONDARY OUTCOMES:
Coma Near Coma Scale | 1 day
  Diagnostic tool for disorders of consciousness. Measuring wakefulness and awareness using sensory stimulation and ratings form responses.
  It is a scale comprised of 11 items with ratings for responses (0, 2, 4; 0 representing higher level response and 4 representing no response). The total score is calculated by adding the ratings and dividing by the number of items scored. Lower numbers indicate greater awareness/consciousness. The ranges are as follows:
  * 0.00-0.89 indicates NO COMA
  * 0.90-2.00 indicates NEAR COMA
  * 2.01-2.89 indicates MODERATE COMA
  * 2.90-3.49 indicates MARKED COMA
  * 3.50-4.00 indicates EXTREME COMA
Nociception Coma Scale | 1 day
  Assessment tool for measuring responses to potentially painful care and/or stimulation of a potentially painful area. It is a scale comprised of 3 items (motor response, verbal response, and facial expression). Ratings consist of 0, 1, 2, 3, with higher ratings indicating higher level responses.The total score is calculated summing the subscores. The total score range is 0-9. A total score equal to or above 4 suggests the presence of pain.

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan W Pool, PhD, Study Director — Anglia Ruskin University
Locations (3):
- United States (2):
  - Children's Healthcare of Atlanta, Atlanta, Georgia
  - Bethany Children's Health Centre, Bethany, Oklahoma
- The Children's Trust, Tadworth, Surrey, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided
Following completion of the study, de-identified, anonymised data (with participant consent) will be available from the corresponding author. Data made available will include individual-level de-identified, anonymised participant data, excluding audio-visual recordings from the MuSICCA sessions.

REFERENCES:
- [Derived] Pool JW, Siegert RJ, Taylor S, Dunford C, Magee W. Evaluating the validity, reliability and clinical utility of the Music therapy Sensory Instrument for Cognition, Consciousness and Awareness (MuSICCA): protocol of a validation study. BMJ Open. 2020 Aug 13;10(8):e039713. doi: 10.1136/bmjopen-2020-039713. PMID 32792456